CLINICAL TRIAL: NCT03835416
Title: Enhanced Protein Intake During Obesity Reduction in Older Male Veterans: Differences in Physical Function and Muscle Quality Responses by Race
Brief Title: Veterans Achieving Weight Loss and Optimizing Resilience-Using Protein
Acronym: VALOR-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E2843-R
Record Dates: First submitted 2019-01-29; First posted 2019-02-08 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Prediabetes; Obesity
Keywords: obesity; prediabetic state; older person; diet, reducing; protein; muscle function
MeSH Terms: conditions — Prediabetic State; Obesity

STUDY DESIGN:
Intervention Model Description: Two-armed Randomized Controlled Trial. Control group follows RDA-level (0.8 g/kg bw/d)protein weight loss diet. Protein follows higher protein (1.4 g/kg bw/d) weight loss diet with balanced protein at each meal.
Who Masked: Outcomes Assessor
Masking Description: Those responsible for outcomes assessment will be blinded from group treatment arm to every extent possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WL-Control (Experimental): 0.8 g protein per kg body weight. Seven servings of whey protein powder (15 g/serving) per week will be provided to participants to support diet affordability.
  Interventions: Dietary Supplement: Foods rich in high quality protein
- WL-Protein (Experimental): >30 g of high quality protein per meal, 1.4 g protein/kg body weight/day. 21 servings of high quality (30 g/serving) protein (lean meats, whey protein powder, protein drinks) provided to participants each week to increase compliance.
  Interventions: Dietary Supplement: Foods rich in high quality protein

INTERVENTIONS:
Dietary Supplement: Foods rich in high quality protein — Along with a weight reduction diet (by instruction), participants will receive high quality protein foods provided to them to include in their daily diet (see study arm description).

SUMMARY:
Diabetes is a major health concern in obese older Veterans, especially in those who are African American. The negative impact of diabetes on muscle and physical function contributes to metabolic as well as physical decline and is under-studied. This randomized controlled trial compares a higher-protein, weight loss regimen previously shown to improve physical function to an Recommended Dietary Allowance (RDA) protein intervention in obese older male Veterans with pre-diabetes and functional limitations. Equal numbers of white and black male Veterans will be studied, filling gaps in the investigators' knowledge of differential responses by race as well as obesity interventions for men in general. The primary outcome is functional performance by Short Physical Performance Battery and secondary measures include muscle quantity and composition, glucose handling, lean body mass, recent falls and fear of falling, and quality of life measured at 0, 3 and 6 months. The goal of this research is to accelerate functional recovery and enhance independence in obese male Veterans, which is strongly aligned with the VA mission to "maximize the physical and social autonomy of Veterans".

DETAILED DESCRIPTION:
This study examines an evidence-based obesity intervention as a means of reducing the impact of prediabetes on muscle function in obese older men of white and black race. A total of 64 obese (BMI 30 kg/m2) male Veterans aged 55 + yrs, with mild to moderate functional impairments (Short Physical Performance Battery score of 4 to 11 units) and prediabetes, will be randomized to a higher-protein weight loss treatment (HP-WL) or an RDA-level protein control weight loss treatment (C-WL). All participants receive individualized calorie prescriptions calculated to achieve a weight loss of ~1-2 pounds per week and attend weekly group support sessions designed to enhance diet compliance with goal setting, self-monitoring, stress management, and daily diet journaling. They will also attend a weekly low impact, chair exercise class. HP-WL participants are provided a supply of chilled/frozen high-quality protein foods (lean meats, low fat dairy products) sufficient to give 30 g high quality protein for two of three meals daily to help assure diet compliance. C-WL participants are provided 1 serving per day of high quality protein to avoid unintentional bias. Treatment responses will be compared for the primary outcome of functional performance by Short Physical Performance Battery and important secondary measures, including muscle quantity and composition, glucose handling, lean body mass, recent falls and fear of falling, and quality of life at 0, 3 and 6 months. An exploratory aim examines potential mediators of racial differences in treatment responses and documents the most successful intervention strategies. This randomized controlled trial of a balanced, higher-protein diet during a metabolic challenge (caloric restriction) in those with prediabetes also considers racial differences in responses of obese older men to this regimen. Study findings will fulfill the RR&D mission by advancing interventions to improve physical function in older Veterans, yield novel information about the impact of balanced, higher protein on muscle and glucose handling, and explore racial differences in responses to obesity interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male Veterans
* African American or Caucasian
* Obese (BMI > 30 kg/m2)
* Age 55+ years
* Pre-diabetes (confirmed fasting plasma glucose 100 and <126 mg/dL) or HbA1c 5.7-6.4%
* Short Physical Performance Battery score of 4 to 11 units
* Age-normal renal function
* English speaking
* Able to record dietary intake or has a proxy who can record dietary intake
* Willing and able to be randomized to either intervention group

Exclusion Criteria:

* Presence of unstable or symptomatic life-threatening illness
* Glomerular filtration rates (GFR) less than 45 mL/min

  * A GFR of 45-59 requires bi-monthly testing per the investigators' established algorithm
  * Those with a GFR <45 mL/min are excluded
* Mini Cog score of <3

  --Vegetarian
* Neurological conditions causing functional impairments, including:

  * Parkinson's Disease
  * multiple sclerosis
  * permanent disability due to stroke
* Inability to complete physical function assessment
* History of significant weight instability
* Contraindicated medications, including narcotic mail-outs and active substance abuse
* Any psychiatric condition that would prevent the subject from participating in a group intervention setting, including diagnosed personality disorders
* Primary care provider disapproves participation

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie W Bales, PhD RD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on medical record queries and letters and at Veteran organizations between September 2019 and October 2023. The first participant was enrolled on 12/12/2019 and the last participant was enrolled on 10/27/2023.
Pre-assignment Details: SPPB and A1c or fasting glucose collected after consent were part of eligibility criteria. Of 105 enrolled participants, 64 met inclusion criteria and were randomized in the trial.
Period: Overall Study
Arm/Group | WL-Control | WL-Protein
Started | 32 | 32
Completed | 20 | 25
Not Completed | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WL-Control | WL-Protein | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (6.9) | 65.9 (6.8) | 67.6 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 32 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 16 | 32
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 32 | 64
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 35.0 (4.2) | 36.5 (4.3) | 35.8 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Total Short Physical Performance Battery (SPPB) Score at Baseline
Description: SPPB total score is the sum of scores from 3 measures, namely balance, gait speed, and chair stands. Score scale 0-12. Higher numbers indicate higher functioning.
Time Frame: 0 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 32 | 32
score on a scale | 9.5 (1.3) | 9.6 (1.2)

2. Primary Outcome: Change in Total Short Physical Performance Battery (SPPB) Score at 3 Months
Description: SPPB total score is the sum of scores from 3 measures, namely balance, gait speed, and chair stands. Score scale 0-12. Higher numbers indicate higher functioning. The change score is determined by the value at 3 months minus the value at baseline.
Time Frame: Baseline and 3 months
Population: A small number of participants do not have this measurement due to COVID-19 disruptions to clinical research, missed appointments, or participant withdrawals/dropouts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 18 | 21
score on a scale | 1.22 (1.17) | 1.48 (1.03)

3. Primary Outcome: Change in Total Short Physical Performance Battery (SPPB) Score at 6 Months
Description: SPPB total score is the sum of scores from 3 measures, namely balance, gait speed, and chair stands. Score scale 0-12. Higher numbers indicate higher functioning. The change score is determined by the value at 6 months minus the value at baseline.
Time Frame: Baseline and 6 months
Population: A small number of participants do not have this measurement due to COVID-19 disruptions to clinical research, missed appointments, or participant withdrawals/dropouts. Additionally, some study participants were enrolled for a 3 month, rather than a 6 month, intervention period, thus they have no measurements at 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 12 | 20
score on a scale | 1.00 (1.28) | 1.85 (1.23)

4. Secondary Outcome: Percent Change in Body Weight at 3 Months
Description: Body weight was measured on the same scale, with light clothing and no shoes, measured to nearest 0.1 lbs. Percent change in body weight was calculated by subtracting weight at 3 months from weight at baseline, dividing by weight at baseline, and multiplying by 100.
Time Frame: Baseline and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in body weight
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 18 | 21
percent change in body weight | -3.1 (3.0) | -4.7 (4.1)

5. Secondary Outcome: Percent Change in Body Weight at 6 Months
Description: Body weight was measured on the same scale, with light clothing and no shoes, measured to nearest 0.1 lbs. Percent change in body weight was calculated by subtracting weight at 6 months from weight at baseline, dividing by weight at baseline, and multiplying by 100.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change of body weight
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 12 | 20
percent change of body weight | -6.5 (4.6) | -6.2 (4.7)

6. Secondary Outcome: Change in 6 Minute Walk Test (Aerobic Endurance) at 3 Months
Description: Meters walked in six minutes on a designated course. Change in meters walked was calculated by subtracting meters walked at 3 months from meters walked at baseline.
Time Frame: Baseline and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 17 | 21
meters | 34.32 (49.10) | 63.29 (58.71)

7. Secondary Outcome: Change in 6 Minute Walk Test (Aerobic Endurance) at 6 Months
Description: Meters walked in six minutes on a designated course. Change in meters walked was calculated by subtracting meters walked at 6 months from meters walked at baseline.
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 12 | 20
meters | 68.10 (39.29) | 65.90 (61.57)

8. Secondary Outcome: Change in Timed 8-ft Up and Go (Agility/Dynamic Balance) at 3 Months
Description: Begins seated. On word 'go' stands, walks around a cone 8 feet away, returns to seated. Timing starts on 'go' and ends when seated. Change in time walked was calculated by subtracting time walked at 3 months from time walked at baseline.
Time Frame: Baseline and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 17 | 21
seconds | -1.58 (1.29) | -1.90 (1.96)

9. Secondary Outcome: Change in Timed 8-ft Up and Go (Agility/Dynamic Balance) at 6 Months
Description: Begins seated. On word 'go' stands, walks around a cone 8 feet away, returns to seated. Timing starts on 'go' and ends when seated. Change in time walked was calculated by subtracting time walked at 6 months from time walked at baseline.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 12 | 20
seconds | -2.10 (0.88) | -2.12 (2.27)

10. Secondary Outcome: Change in Number of Chair Stands in 30 Seconds (Lower Body Strength) at 3 Months
Description: With arms across chest, stand up completely and return to seated as many times as possible in 30 seconds. Change in number of chair stands was calculated by subtracting number of chair stands at 3 months from number of chair stands at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

11. Secondary Outcome: Change in Number of Chair Stands in 30 Seconds (Lower Body Strength) at 6 Months
Description: With arms across chest, stand up completely and return to seated as many times as possible in 30 seconds. Change in number of chair stands was calculated by subtracting number of chair stands at 6 months from number of chair stands at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

12. Secondary Outcome: Change in Isokinetic Knee Extension Peak Torque (Muscle Strength) at 3 Months
Description: Knee extensor at 60 degrees with a dynamometer. Average peak torque for three trials will be recorded. Change in peak torque was calculated by subtracting peak torque at 3 months from peak torque at baseline.
Time Frame: Baseline and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: newton-meters
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 17 | 21
newton-meters | -5.02 (20.65) | 4.66 (31.54)

13. Secondary Outcome: Change in Isokinetic Knee Extension Peak Torque (Muscle Strength) at 6 Months
Description: Knee extensor at 60 degrees with a dynamometer. Average peak torque for three trials will be recorded. Change in peak torque was calculated by subtracting peak torque at 6 months from peak torque at baseline.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: newton-meters
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 12 | 20
newton-meters | -7.20 (18.92) | -3.98 (33.50)

14. Secondary Outcome: Change in Isometric Hand Grip (Upper Body Strength) at 3 Months
Description: Using the Jamar Hand Dynamometer, the amount of pressure placed when squeezing the instrument as hard as possible was measured. Two trials per hand were measured. Change in hand grip was calculated by subtracting the highest value at 3 months from the highest value at baseline.
Time Frame: Baseline and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 18 | 21
kilograms | 0.85 (4.32) | 3.69 (5.61)

15. Secondary Outcome: Change in Isometric Hand Grip (Upper Body Strength) at 6 Months
Description: Using the Jamar Hand Dynamometer, the amount of pressure placed when squeezing the instrument as hard as possible was measured. Two trials per hand were measured. Change in hand grip was calculated by subtracting the highest value at 6 months from the highest value at baseline.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 12 | 20
kilograms | 1.21 (5.02) | 3.01 (6.55)

16. Secondary Outcome: Change in Minimal Waist Circumference at 3 Months
Description: Minimal waist circumference was measured at smallest horizontal circumference above umbilicus and below xiphoid process. Change in minimal waist circumference was calculated by subtracting the measurement at 3 months from the measurement at baseline.
Time Frame: Baseline and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 18 | 21
centimeters | -2.64 (3.76) | -4.12 (3.90)

17. Secondary Outcome: Change in Minimal Waist Circumference at 6 Months
Description: Minimal waist circumference was measured at smallest horizontal circumference above umbilicus and below xiphoid process. Change in minimal waist circumference was calculated by subtracting the measurement at 6 months from the measurement at baseline.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 12 | 20
centimeters | -4.95 (5.10) | -4.81 (4.30)

18. Secondary Outcome: Change in Body Composition: Percent Lean Mass at 3 Months
Description: Air displacement plethysmography method (Life Measurement, Inc., Concord, CA). The Cardio Pulmonary, Metabolic and Body Composition (COSMED) BodPod has excellent sensitivity and test-to-test reliability, ease of use, and non-invasive nature, which is important for full participation from this population. Percent lean mass was calculated by the BodPod machine and entered into a REDCap database. Then, change in percent lean mass was calculated by subtracting the percent lean mass at 3 months from the percent lean mass at baseline.
Time Frame: Baseline and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change in total lean mass percentage
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 18 | 21
change in total lean mass percentage | 1.11 (1.57) | 2.37 (2.37)

19. Secondary Outcome: Change in Body Composition: Percent Lean Mass at 6 Months
Description: Air displacement plethysmography method (Life Measurement, Inc., Concord, CA). The Cardio Pulmonary, Metabolic and Body Composition (COSMED) BodPod has excellent sensitivity and test-to-test reliability, ease of use, and non-invasive nature, which is important for full participation from this population. Percent lean mass was calculated by the BodPod machine and entered into a REDCap database. Then, change in percent lean mass was calculated by subtracting the percent lean mass at 6 months from the percent lean mass at baseline.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: change in total lean mass percentage
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 12 | 20
change in total lean mass percentage | 2.95 (2.94) | 3.31 (2.77)

20. Secondary Outcome: Change in Body Composition: Percent Fat Mass at 3 Months
Description: Air displacement plethysmography method (Life Measurement, Inc., Concord, CA). The Cardio Pulmonary, Metabolic and Body Composition (COSMED) BodPod has excellent sensitivity and test-to-test reliability, ease of use, and non-invasive nature, which is important for full participation from this population. Percent fat mass was calculated by the BodPod machine and entered into a REDCap database. Then, change in percent fat mass was calculated by subtracting the percent fat mass at 3 months from the percent fat mass at baseline.
Time Frame: Baseline and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change in total body fat mass percentage
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 18 | 21
change in total body fat mass percentage | -1.11 (1.57) | -2.37 (2.37)

21. Secondary Outcome: Change in Body Composition: Percent Fat Mass at 6 Months
Description: Air displacement plethysmography method (Life Measurement, Inc., Concord, CA). The Cardio Pulmonary, Metabolic and Body Composition (COSMED) BodPod has excellent sensitivity and test-to-test reliability, ease of use, and non-invasive nature, which is important for full participation from this population. Percent fat mass was calculated by the BodPod machine and entered into a REDCap database. Then, change in percent fat mass was calculated by subtracting the percent fat mass at 6 months from the percent fat mass at baseline.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: change in total body fat mass percentage
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 12 | 20
change in total body fat mass percentage | -2.95 (2.94) | -3.31 (2.77)

22. Secondary Outcome: Mini-Cog at Baseline Only
Description: To assess for cognitive impairment, the mini cog was used to screen for eligibility at baseline only. The mini cog includes two components - a 3-item recall and a clock drawing. You can score 0-3 points for the 3-item recall, and 0-2 points for the clock drawing. These subscale scores are summed for a total possible score of 5. Subscale scores were not reported, only the total score. The total score is a range of 0-5. The max total score is 5 with 5 being the best score. To be eligible for the study, the total item recall and clock score needed to be 3 or higher.
Time Frame: Baseline only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 32 | 32
score on a scale | 3.97 (0.90) | 4.06 (0.98)

23. Secondary Outcome: Change in Computerized Axial Tomography (CAT) Scan at 3 Months
Description: Cross sectional area of the thigh to determine thigh muscle mass. Change in area calculated by subtracting area at 3 months from area at baseline.
Time Frame: Baseline and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 22 | 19
cm^2 | 1.68 (16.79) | 4.65 (18.76)

24. Secondary Outcome: Change in Computerized Axial Tomography (CAT) Scan at 6 Months
Description: Cross sectional area of the thigh to determine thigh muscle mass. Change in area calculated by subtracting area at 6 Months from area at baseline.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 14 | 10
cm^2 | 7.22 (22.20) | 2.43 (13.95)

25. Secondary Outcome: Change in Short Form-36 (SF-36) Health Survey at 3 Months
Description: Quality of Life Questionnaires The SF-36 measures 8 QOL domains which are dichotomized into physical (functioning, role limitations-physical, pain, general health) and mental health (vitality, social functioning, role limitations-emotional, and emotional/mental health). Item scores were converted to a 0-100 point scale; domain scores were derived by averaging individual items within the subscale; and physical composite and mental health composite scores were derived by averaging the four component domains of each. Higher values are indicative of better QOL. Change in score calculated by subtracting score at 3 months from score at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

26. Secondary Outcome: Change in Short Form-36 (SF-36) Health Survey at 6 Months
Description: Quality of Life Questionnaires The SF-36 measures 8 QOL domains which are dichotomized into physical (functioning, role limitations-physical, pain, general health) and mental health (vitality, social functioning, role limitations-emotional, and emotional/mental health). Item scores were converted to a 0-100 point scale; domain scores were derived by averaging individual items within the subscale; and physical composite and mental health composite scores were derived by averaging the four component domains of each. Higher values are indicative of better QOL. Change in score calculated by subtracting score at 6 months from score at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

27. Secondary Outcome: Change in Profile of Mood States (POMS) at 3 Months
Description: Mood Questionnaires The 30-item POMS measures mood and mood changes, has low respondent burden, and includes 6 subscales: tension, depression, anger, fatigue, confusion and vigor (all with range 0-20). Total mood disturbance (TMD) is derived from POMS using the following formula, TMD = (Sum of all subscales except vigor) - vigor (range -20 - 100). Change in score calculated by subtracting score at 3 months from score at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

28. Secondary Outcome: Change in Profile of Mood States (POMS) at 6 Months
Description: Mood Questionnaires The 30-item POMS measures mood and mood changes, has low respondent burden, and includes 6 subscales: tension, depression, anger, fatigue, confusion and vigor (all with range 0-20). Total mood disturbance (TMD) is derived from POMS using the following formula, TMD = (Sum of all subscales except vigor) - vigor (range -20 - 100). Change in score calculated by subtracting score at 6 months from score at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

29. Secondary Outcome: Change in Center for Epidemiologic Studies Depression Scale (CES-D) at 3 Months
Description: Depression Questionnaires Individuals were coded as positive for depression if they had a CES-D score of 16 and/or had self-report of depression diagnosis at baseline. In addition to the total score, the CES-D includes 4 subscales: depressed affect (range 0-21), positive affect (range 0-12), somatic (range 0-21), and interpersonal (range 0-6). Change in score calculated by subtracting score at 3 months from score at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

30. Secondary Outcome: Change in Center for Epidemiologic Studies Depression Scale (CES-D) at 6 Months
Description: Depression Questionnaires Individuals were coded as positive for depression if they had a CES-D score of 16 and/or had self-report of depression diagnosis at baseline. In addition to the total score, the CES-D includes 4 subscales: depressed affect (range 0-21), positive affect (range 0-12), somatic (range 0-21), and interpersonal (range 0-6). Change in score calculated by subtracting score at 6 months from score at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

31. Secondary Outcome: Change in Perceived Stress Scale (PSS) at 3 Months
Description: Stress Questionnaires The PSS assesses the degree to which situations in one's life are considered stressful (range 0-40).
  Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
  Change in score calculated by subtracting score at 3 months from score at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

32. Secondary Outcome: Change in Perceived Stress Scale (PSS) at 6 Months
Description: Stress Questionnaires The PSS assesses the degree to which situations in one's life are considered stressful (range 0-40).
  Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
  Change in score calculated by subtracting score at 6 months from score at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

33. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) and 3 Months
Description: Quality of sleep Questionnaires Reported PSQI values include only these six component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, and use of sleeping medication (all with a range 0-3).
  The PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
  Change in score calculated by subtracting score at 3 months from score at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

34. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) and 6 Months
Description: Quality of sleep Questionnaires Reported PSQI values include only these six component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, and use of sleeping medication (all with a range 0-3).
  The PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality. Change in score calculated by subtracting score at 6 months from score at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

35. Secondary Outcome: Change in Satisfaction With Life Scale (SWLS) at 3 Months
Description: Life Satisfaction Questionnaires The SWLS evaluates global life satisfaction, an important component of subjective well-being (range 5-35).
  The SWLS is a 7-point Likert scale style response scale. The possible range of scores is 5-35, with a score of 20 representing a neutral point on the scale. Scores between 5-9 indicate the respondent is extremely dissatisfied with life, whereas scores between 31-35 indicate the respondent is extremely satisfied. Change in score calculated by subtracting score at 3 months from score at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

36. Secondary Outcome: Change in Satisfaction With Life Scale (SWLS) at 6 Months
Description: Life Satisfaction Questionnaires The SWLS evaluates global life satisfaction, an important component of subjective well-being (range 5-35).
  The SWLS is a 7-point Likert scale style response scale. The possible range of scores is 5-35, with a score of 20 representing a neutral point on the scale. Scores between 5-9 indicate the respondent is extremely dissatisfied with life, whereas scores between 31-35 indicate the respondent is extremely satisfied. Change in score calculated by subtracting score at 6 months from score at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

37. Secondary Outcome: Change in Hemoglobin A1c at 3 Months
Description: Blood assay (LabCorp). Change in value calculated by subtracting value at 3 months from value at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

38. Secondary Outcome: Change in Hemoglobin A1c at 6 Months
Description: Blood assay (LabCorp). Change in value calculated by subtracting value at 6 months from value at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

39. Secondary Outcome: Change in Fear of Falling at 3 Months
Description: "Yes" responses to the question, "Do you have a fear of falling?" Change in number of "yes" answers from baseline to 3 months. Change was calculated by subtracting the number of "yes" answers at 3 months from the number of "yes" answers at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

40. Secondary Outcome: Change in Fear of Falling at 6 Months
Description: "Yes" responses to the question, "Do you have a fear of falling?" Change in number of "yes" answers from baseline to 6 months. Change was calculated by subtracting the number of "yes" answers at 6 months from the number of "yes" answers at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

41. Secondary Outcome: Change in Number of Falls at 3 Months
Description: This is an open-ended questionnaire to see the change in number of times a person falls between time points. Change in value calculated by subtracting value at 3 months from value at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

42. Secondary Outcome: Change in Number of Falls at 6 Months
Description: This is an open-ended questionnaire to see the change in number of times a person falls between time points. Change in value calculated by subtracting value at 6 months from value at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

43. Secondary Outcome: Change in 3-day Diet Record, Calories, at 3 Months
Description: 3-day diet record by multiple pass; analyzed Food Processor (Version 10.13, 2013; ESHA Research). Change in calories calculated by subtracting average daily calories at 3 months from average daily calories at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

44. Secondary Outcome: Change in 3-day Diet Record, Calories, at 6 Months
Description: 3-day diet record by multiple pass; analyzed Food Processor (Version 10.13, 2013; ESHA Research). Change in calories calculated by subtracting average daily calories at 6 months from average daily calories at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

45. Secondary Outcome: Change in 3-day Diet Record, Protein, at 3 Months
Description: 3-day diet record by multiple pass; analyzed Food Processor (Version 10.13, 2013; ESHA Research). Change in protein in grams calculated by subtracting average daily protein in grams at 3 months from average daily protein in grams at baseline.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

46. Secondary Outcome: Change in 3-day Diet Record, Protein, at 6 Months
Description: 3-day diet record by multiple pass; analyzed Food Processor (Version 10.13, 2013; ESHA Research). Change in protein in grams calculated by subtracting average daily protein in grams at 6 months from average daily protein in grams at baseline.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

47. Secondary Outcome: Number of Participants Measured Using an Axis Accelerometer (Actigraph)
Description: Actigraph WGT3X-BT is a wearable accelerometer that measures activity counts, step counts, and physical activity intensity. This outcome is the number of participants who participated in this measurement at baseline.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 32 | 32
Participants | 32 | 32

48. Secondary Outcome: Number of Participants Measured Using an Axis Accelerometer (Actigraph)
Description: Actigraph WGT3X-BT is a wearable accelerometer that measures activity counts, step counts, and physical activity intensity. This outcome is the number of participants who participated in this measurement at 3 months.
Time Frame: 3 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 32 | 32
Participants | 17 | 21

49. Secondary Outcome: Number of Participants Measured Using an Axis Accelerometer (Actigraph)
Description: Actigraph WGT3X-BT is a wearable accelerometer that measures activity counts, step counts, and physical activity intensity. This outcome is the number of participants who participated in this measurement at 6 months.
Time Frame: 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 32 | 32
Participants | 12 | 20

50. Secondary Outcome: Change in Glucose Tolerance Test (OGTT) (78-80), Blood
Description: Ingestion of a 75 g glucose load
Time Frame: 3 months
Population: These data were unable to be collected due to methodologic difficulties and logistical constraints.
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: Change in Glucose Tolerance Test (OGTT) (78-80), Blood
Description: Ingestion of a 75 g glucose load
Time Frame: 6 months
Population: These data were unable to be collected due to methodologic difficulties and logistical constraints.
Arm/Group | WL-Control | WL-Protein
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: Percent Attendance at Weekly Diet Class Between Baseline and 3 Months
Description: Attendance counted if in person or virtual. Percentage calculated by dividing number of classes attended by number of classes held and multiplying by 100.
Time Frame: Baseline and 3 months
Reporting Status: Not Posted, anticipated posting 2026-03

53. Secondary Outcome: Percent Attendance at Weekly Diet Class Between Baseline and 6 Months
Description: as for outcome 52
Time Frame: Baseline and 6 months
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: From time of consent to completion of either 3 month or 6 month study, 4-7 months
Groups:
- Consented, Not Randomized: Participants who consented but were never randomized due to participant withdrawal or not qualifying.
Arm/Group | WL-Control | WL-Protein | Consented, Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/32 | 1/32 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/32 | 0/41
Other Adverse Events (participants affected / at risk) | 10/32 | 13/32 | 2/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WL-Control (N=32) | WL-Protein (N=32) | Consented, Not Randomized (N=41)
Death (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WL-Control (N=32) | WL-Protein (N=32) | Consented, Not Randomized (N=41)
Bladder tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — Identified while in study
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0
Surgery (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Removal of melanoma
Broken bone (Injury, poisoning and procedural complications) | 0 | 2 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal Stenosis (Surgical and medical procedures) | 0 | 1 | 0
Complications from Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (2) | 0 — Pre-existing condition
Frequent Urination (Renal and urinary disorders) | 0 | 1 | 0
Respiratory Illness (Infections and infestations) | 3 | 1 | 0
Dizziness, nausea, abdominal pain (General disorders) | 0 | 2 | 1
Shoulder pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Adrenal gland removal (Surgical and medical procedures) | 0 | 0 | 1
Shoulder surgery (Surgical and medical procedures) | 1 | 0 | 0 — Due to prior injury
Eye pain (Eye disorders) | 0 | 1 | 0 — Due to past injury.
Leg pain/weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — Attributed to arthritis
Elevated blood pressure (Vascular disorders) | 1 | 1 | 0
ED visit for difficulty breathing/coughing blood possibly related to congestive heart failure (General disorders) | 1 | 0 | 0
Shingles (Infections and infestations) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bursitis in elbow (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood clot in eye (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gluteal cleft abscess (Infections and infestations) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
The outcomes for which data are missing have the following explanations:

1. Data were collected but the data analysis is still in progress.
2. We were unable to collect the outcome due to financial and logistical restrictions or the inability to establish satisfactory sample collection processes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT03835416/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT03835416/ICF_000.pdf